# **RESEARCH PROTOCOL**

# **Protocol Title and Number:**

A randomized trial of a text message quit vaping intervention for young adults

## **Date of Submission to Advarra:**

May 28, 2020

# Sponsor:

Truth Initiative 900 G Street, NW Fourth Floor Washington, DC 20001

# **Principal Investigator:**

Amanda L. Graham, PhD Chief, Innovations Truth Initiative 900 G Street, NW Fourth Floor Washington, DC 20001

T: 202/454-5938

agraham@truthinitiative.org

# **Final Signed Protocol:**

Amanda L. Graham, PhD

Principal Investigator Name

Principal Investigator Signature

Amandol Eraham

May 28, 2020

Date

#### **BACKGROUND**

The popularity of electronic cigarettes (or e-cigarettes) has grown exponentially over the past few years, with the surgeon general calling the use of e-cigarettes among young people an "epidemic". E-cigarettes are now the most commonly used tobacco product among youth and in the U.S., youth and young adults are more likely than adults to use e-cigarettes. Many younger e-cigarette users have never used another tobacco product: among current e-cigarette users aged 45 years and older in 2015, most were either current or former regular cigarette smokers; in contrast, among current e-cigarette users aged 18-24 years, 40.0% had never been regular cigarette smokers. E-cigarette use has grown even faster in recent years due to the popularity of products such as

JUUL, a small-USB like e-cigarette with high nicotine content that is easy to conceal. A 2018 study by our colleagues at Truth Initiative showed that the highest percentage of e-cigarette users were ages 18-21 years old.<sup>3</sup>

Young people should never use nicotine in any form. While there is some evidence that e-cigarettes are less harmful than traditional cigarettes, they are not harmless and early exposure to nicotine can have long-lasting adverse effects. The majority of e-cigarettes contain nicotine, which has known health effects on brain development which occurs



into the mid-20s. Specific risks include nicotine addiction, mood disorders, permanent lowering of impulse control, as well as negative impacts on attention and learning. The aerosol produced by e-cigarettes contains cancer-causing chemicals and tiny particles that reach deep into the lungs. E-cigarettes have also produced unintended injuries such as fires and explosions from defective batteries and poisonings from acute nicotine exposure through e-cigarette liquids. Finally, there is strong evidence that e-cigarette use can lead to the use of other tobacco products such as cigarettes.<sup>4,5</sup> Reversing the dramatic gains over the past decade in reducing cigarette smoking among young people would be nothing short of a public health tragedy.

In response to this epidemic and given no available quitting resources for young people (cessation resources such as medication have no demonstrated effectiveness for young people<sup>6,7</sup>), Truth Initiative launched a first-of-its kind e-cigarette cessation program designed specifically for young people in January 2019. The program is called *This is Quitting* and it is delivered entirely via text message. Mobile phone ownership is ubiquitous among young people and text messaging is a preferred communication modality in this age group. Text messaging is also easy to use, discreet, anonymous, and there is strong evidence supporting its effectiveness as a cessation intervention modality. *This is Quitting* was developed using best practices from smoking cessation research with young people, our extensive experience delivering digital tobacco cessation interventions to people of all ages, as well as formative research with young e-cigarette users and quitters.

Young people enroll by texting "DITCHJUUL" to a short code and responding to the initial message with their age and first name (used for tailoring the program). Terms of Service and Privacy Policy are provided via a link in a text message (included in Appendix A). Users receive one age-appropriate message per day tailored to their enrollment date or quit date, which can be set and reset via text message. Those not ready to quit receive 4 weeks of messages focused on building skills and confidence. Users who set a quit date receive messages for a week preceding it and 8 weeks afterward that include encouragement and support, skill- and self-efficacy building exercises, coping strategies, and information about the risks of vaping, benefits of quitting, and cutting down to quit. Keywords COPE, STRESS, SLIP, and MORE provide on-demand support. Sample text messages can be found at the end of this protocol. Users can unsubscribe anytime by texting STOP. E-cigarette use and abstinence are assessed via text message at 14, 30, 60, and 90 days following an enrollee's quit date or enrollment date. At 14 days, enrollees are asked, "Have you cut down how much you JUUL in the past 2 weeks? Respond w/letter: A=I still JUUL the same amount, B=I JUUL less, C=I don't JUUL at all anymore." At 30, 60, and 90 days, enrollees are asked, "When was the last time you JUULed, even a puff of someone else's? Respond w/ letter: A: in the past 7 days, B: 8–30 days ago, C: More than 30 days ago."

To date, more than <u>58,000 young people have enrolled</u>, demonstrating the appeal of this treatment approach and the urgent need for quit vaping resources among young people. Preliminary evaluation data collected among an initial cohort of roughly 27,000 users has shown high levels of engagement in the program and high rates of abstinence among responders. Roughly 4 of users set a quit date, with the most common quit date being the day of enrollment. Interactive keywords were used by 45.5% of teens and 38.4% of YA. Response rates to follow-up assessment questions were 36.9% at 14 days and 21.0% at 90 days. At 14 days, 60.8% of respondents indicated they had reduced or stopped using e-cigarettes altogether. At 90 days, 7-day point prevalence abstinence (ppa) was 25% and 30-day ppa was 16%. The high volume of enrollment in a short period of time, high levels of

engagement with the program, and e-cigarette reduction and cessation results demonstrate that young people are interested in quitting vaping and can be engaged in an easily accessible, anonymous digital platform.

Building on this preliminary evidence, the primary aim of the current study is to conduct a fully powered comparative effectiveness trial to evaluate the effectiveness of *This is Quitting* in promoting abstinence from e-cigarettes among young users aged 18-24. This study is a 2-arm randomized controlled trial conducted among young users aged 18-24 recruited through online channels. Participants will be randomized to *This is Quitting* or to an assessment-only control condition and followed for 7 months to roughly correspond to 6-months post-treatment. The secondary aim is to examine potential mediators of program effectiveness, including treatment engagement and changes in self-efficacy and perceived social support for quitting.

The scientific, clinical, and public health communities are desperate for proven, evidence-based cessation resources to address the vaping epidemic among young people. We are uniquely positioned to address this urgent need given our extensive experience in conducting large-scale, rigorous research trials of digital tobacco cessation interventions and our expertise in working with young people. We plan to rapidly disseminate study results to benefit other researchers/service providers and use these results to further enhance the program.

#### **METHODS**

## **Subjects**

We will recruit N=2600 e-cigarette users aged 18-24 years old who are interested in quitting in the next 30 days. Other eligibility criteria include past 30-day e-cigarette use and US residence. To fully enroll in the study, individuals must sign up for *This is Quitting* and respond to the initial system-generated message.

#### **Recruitment and Enrollment**

Potential participants will respond to online ads on various platforms (Facebook, YouTube, Instagram, Reddit, etc.) if they are current e-cigarette users who are interested in quitting and willing to participate in a research study. Clicking on the ad will lead them to a webpage that provides details about what participation in the study entails and describes incentives for participation. Those who are interested will complete an eligibility screener followed by informed consent and a baseline assessment. Those who complete the baseline will be randomized into one of two arms (see below for additional details) and instructed to text a specific keyword to the phone number corresponding to their treatment assignment. Only those who respond to the first message from the text message program within 24 hours will be fully enrolled into the study. This requirement will be made explicit.

#### Randomization

Randomization occurs after completion of the online enrollment process (completed baseline survey). A computer algorithm that is part of the survey software will automate random allocation.

#### Interventions

**This is Quitting:** Participants will be enrolled to receive messages from This is Quitting as described above. **Assessment-only control.** After an initial enrollment message, participants will be contacted periodically to assess e-cigarette use. At the end of the intervention period, they will receive information on how to sign up for This is Quitting if they are interested in the program (optional).

# **Potential Problems and Solutions**

Loss to follow-up is the primary concern in trials involving digital interventions, especially ones that employ an assessment only control. We expect at least 75% follow-up at 1-month and 65% at 7-months based on our previous and ongoing digital mobile-based evaluations. If follow-up rates are lower than expected early in the trial, we will consider shortening the 7-month follow-up to gather only abstinence outcomes. To maximize follow up rates we will:

- 1) provide clear information about the study at the outset, including expectations for follow-up;
- 2) reimburse participants up to \$30 per follow-up assessment;
- 3) collect interim abstinence assessments via text (\$5 incentive for each response) for both arms to optimize the likelihood that participants randomized to the assessment-only control stay engaged with the study;
- 4) send reminders about follow-up surveys via email and text messages;
- 5) conduct phone follow-ups for those unreachable by email and text messages; and,

6) emphasize the importance of survey completion regardless of abstinence status.

#### Measures

All randomized participants in both arms will be asked to complete all assessments. Assessments will occur at baseline and 1 month and 7 months post-randomization. The baseline survey will be conducted online and hosted on a secure server. Mixed-mode follow-up (email, phone, text) will be employed. Telephone surveys will be conducted by research staff blind to treatment. Text messages have demonstrated moderately high reliability (k=.66) compared with web-based surveys in assessing smoking outcomes<sup>10</sup> and will be used as a final means of gathering abstinence data from non-responders. Most measures listed below are standard instruments used in cessation studies, and are reliable when administered via the Internet.<sup>11,12</sup>

**Screening Variables.** To characterize the sample of users interested in the study and assess for eligibility, we will gather: <u>demographics</u> (age, education, income level, sexual and gender identity, race, and ethnicity); <u>current e-cigarette use</u> (use of e-cigarette containing nicotine or THC in the past 30 days)<sup>13</sup>; <u>interest in quitting</u>; <u>contact information</u> (e-mail and phone number to send baseline survey to and link text message sign-up data). These questions are being asked up front so we can determine whether users enrolling in the study are representative of the wider population of e-cigarette users.

**Baseline Variables.** To characterize the sample and explore potential moderators of treatment effectiveness, we will gather: additional <u>demographics</u> (student status, employment status); <u>current e-cigarette use and history</u> (frequency and rate, <sup>13,14</sup> motivation to quit and quitting history <sup>15</sup>); <u>nicotine dependence</u> will be assessed with the PROMISE-E<sup>16</sup> and items from the Texas Adolescent and Tobacco Marketing Surveillance <sup>17</sup>; <u>other substance use</u> (other tobacco products, alcohol) <sup>18</sup> and <u>mental health symptoms</u>. <sup>19</sup> Given evolving trends of e-cigarette use and perception, we will also ask about their awareness about media reports about e-cigarettes, perception about e-cigarettes, reasons for wanting to quit, and reasons for joining the study. To account for potential predictors of dropout, we will ask about motivation to use or quit e-cigarettes and potential barriers to quitting (e.g., social influences). We will assess baseline levels of perceived level of social support, perceived social norms, and perceived self-efficacy for quitting and examine changes in these variables as potential mediators of treatment effectiveness.

**Mediating Variables.** We hypothesize that treatment engagement will mediate the relationship between treatment assignment and abstinence outcomes. We will extract data regarding replies to interactive text messages (e.g., setting a quit date, keyword use) as well as unsubscribe status, number of days enrolled, and total number of messages received. All text message interactions are date/time stamped.

**Outcome Measures.** The <u>primary outcome</u> is self-reported 30-day point-prevalence abstinence (ppa) at 7-months but we will gather abstinence data at all follow-ups. <u>Other quitting-related outcomes</u> include change in motivation to quit, quit attempts, reduction in e-cigarette use, 7-day ppa, and continuous abstinence measured at each formal follow-up as well as interim text message assessments (single item asking about current vaping status). <u>Intervention satisfaction</u> in both conditions will be measured with items about overall satisfaction and whether they would recommend it to a friend (scale from 0-10). Satisfaction with frequency of text messages will be measured.<sup>20</sup> To assess <u>perceived message relevance</u>, participants will be asked whether text messages "were written personally for you"<sup>21</sup> and "were directed at you personally".<sup>22</sup> Since the intervention is freely available throughout the U.S. through the well-known **truth** campaign, we want to understand the potential impact of <u>brand awareness</u> on engagement with the intervention and outcomes. At the final 7-month follow-up, we will ask a series of questions to establish awareness of the **truth** brand and awareness of This is Quitting among control arm participants. The 7-month follow-up assessment will also be occurring during the unprecedented global health event of COVID-19, so we will be asking questions to assess the <u>impact of COVID-19</u> on the perceptions and behaviors related to vaping to measure any potential impact.

Following the completion of the final 7-month follow-up assessment, after participants receive compensation for completing this survey, we will administer an exit questionnaire that queries participants about the accuracy of their self-reports. This process was used successfully by Lantini et al<sup>23</sup> to determine rates of misreporting of outcomes in a randomized trial with adolescent smokers. Items will address the reasons for joining the study, the extent to which they paid attention to the study questions and their answers, the extent to which they like/dislike the way vaping makes them look, concerns about confidentiality in the study, and several items tapping social desirability bias in the context of a digital intervention.

## **Data Analysis Plan**

**Primary Analysis.** Point-prevalence abstinence (ppa) at 6-months post-treatment will be compared across the treatment and control groups using logistic regression. All estimates will be adjusted for baseline confounders of the intervention-outcome relationship. We will identify potential moderators (e.g., age, gender, baseline motivation to quit) by analyzing interactions

between treatment and selected variables. For all moderators found to be associated with the primary outcome, we will examine the effects of treatment/moderator interaction terms on outcomes after entering main effects.

**Secondary Analyses.** Additional outcomes related to abstinence and treatment engagement will also be analyzed with logistic regression as secondary analyses. These include likelihood of making a quit attempt, likelihood of reducing e-cigarette use, and changes in confidence and self-efficacy in quitting e-cigarettes.

Missing Data. Missing data will be handled in two ways. First, we will conduct an intent-to-treat (ITT) analysis in which participants who have been lost to follow up are assumed to be treatment failures (i.e., vaping). This analysis will be conducted

because ITT analyses are common in the smoking cessation literature, despite simulations demonstrating that the approach is neither conservative nor anticonservative but rather biased in favor of whichever condition contains less missingness. <sup>24</sup> Second, we will supplement the ITT analyses with an analysis that uses a multiple imputation (MI) procedure to minimize bias in estimates and standard errors, under the assumption that outcomes are not missing at random (NMAR) but rather more likely to be missing for treatment failures (i.e., vaping) than treatment successes (i.e. abstinence). Since the magnitude of actual response bias is unknown, we will conduct a sensitivity analysis to evaluate the treatment effect on outcomes under a range of magnitudes, from equal odds of missing (OR=1) to five times more likely to be missing (OR=5).

**Mediator Analysis.** Our conceptual model is that treatment increases the odds of abstinence by increasing perceived social support and perceived self-efficacy for quitting. Those two constructs will be measured at baseline, 1-month and 7-



months post-treatment. Change in those constructs from baseline will be evaluated with separate mediation analyses as presented in Figure 1. Specifically, we hypothesize that the effect of treatment on abstinence will be mediated by perceived social support and perceived self-efficacy, such that: (1) a significant effect A is found associating X with Z; (2) a significant effect B is found associating Z with Y; (3) a significant effect C is found associating X with Y; and (4) the effect of C is significantly attenuated when A and B are simultaneously included in the model.

## **PROTECTION OF HUMAN SUBJECTS**

#### Human Subjects Involvement, Characteristics, and Design

Participants will be 1,720 e-cigarette users aged 18-24 who respond to online advertising about a research study and who complete enrollment into a text message program based on random allocation. Study enrollment is conducted entirely online and is fully automated. Randomization occurs after participants have provided informed consent and completed the baseline survey. Study enrollment will not be considered complete until the participant responds to the initial system-generated text message. There will be no involvement of vulnerable populations and no deception. Children (under the age of 18) will be excluded.

#### **Sources of Materials**

Sources of research material include the following: 1) screening data, 2) text message utilization data, and 3) baseline and follow-up assessments. The baseline assessment will be conducted online with the survey hosted on a secure server. Mixed-mode follow-up (online, phone, text message) will be employed. Phone surveys will be conducted by research staff blind to treatment condition.

#### **Materials Access**

For all data, the Principal Investigator (Dr. Amanda Graham), Data Analyst (Dr. Michael Amato), Project Managers (Sarah Cha, Megan Jacobs), research assistants (Mia Bottcher, Jenna Woodward), and the software development team will have access to individually identifiable information about human subjects. Electronic data files with identifiable information will be maintained separately from other data files and will only be used for administrative purposes (e.g., tracking follow-up completion, managing subject payment). All personnel already have or will have received certification in human subjects protection prior to beginning work on this project.

#### **Potential Risks**

The overall risk is judged to be very low. Study participants who attempt to quit e-cigarette use will likely experience some nicotine withdrawal symptoms that may include anxiety, restlessness, anger, irritability, sadness, and problems concentrating. There is no

reason to believe that participation in this study would worsen nicotine withdrawal symptoms or that symptoms would differ based on randomization assignment.

#### **ADEQUACY OF PROTECTION AGAINST RISKS**

## **Enrollment and Informed Consent**

Step 1 (Study information): Potential participants who click on an online ad for e-cigarette users who are interested in quitting and willing to participate in a research study will be directed to a website that provide additional details about the study. This webpage will provide information on who is behind the study, what participation entails, and who may be eligible for the study. Step 2 (Eligibility screening): Individuals who are interested in participating will complete a short survey to confirm eligibility for study participation. Those who are eligible will be asked to provide contact information (e-mail address to send links to surveys and mobile number for text message sign up). Step 3 (E-mail confirmation): An email message is sent to the participant with a distinct URL (Web address) containing the baseline survey and instructions to complete the survey within 24 hours to complete study enrollment. This process ensures that enrolled participants have a valid email address where they can receive study-related correspondence. Step 4 (Informed consent and baseline assessment): When the participant clicks on the URL in the email, it will open up an online baseline survey. On the first page of the baseline survey, a full informed consent text will be provided, including a) each study condition; b) financial incentives for participating; c) the process of randomization and the equal chance of being assigned to one of two treatment conditions; d) protection of confidentiality and the right to withdraw at any time; and e) expectations regarding follow-up data collection, including compensation for time required to complete follow-up assessments (regardless of e-cigarette use status). Users will be required to select "Yes, I would like to continue" as active affirmation that they are providing informed consent for study participation. Contact information for the study and the Institutional Review Board where IRB approval has been obtained will be included in the consent form. All information about the study will be written at a 6th grade reading level to ensure adequate comprehension. Agreeing to participate will launch the baseline assessment. Step 5 (Randomization): Randomization will only occur after an eligible study participant has completed the online enrollment process (confirmed eligibility, indicated informed consent, and completed baseline survey). Step 6 (Text message sign-up): Users will be randomized at the conclusion of the baseline assessment and provided with a phone number to text based on their assignment. Users must text their assigned number and reply to the welcome text message to confirm text message enrollment and finalize their study enrollment.

#### **Protections Against Risk**

Exposure to evidence-based information and support for e-cigarette cessation in the intervention arm is expected to attenuate withdrawal symptoms associated with e-cigarette cessation that may occur.

# POTENTIAL BENEFITS OF THE PROPOSED RESEARCH TO HUMAN SUBJECTS AND OTHERS

Subjects may benefit from participation in this research in several ways. By participating in an e-cigarette cessation treatment program, subjects may increase the likelihood that they will attempt to quit e-cigarette use and be successful. Alternatively, participants will gain a greater understanding of their e-cigarette use behavior that may help them to quit successfully in the future. Finally, although this is not a direct benefit, all participants will be involved in a project to evaluate innovative treatments for e-cigarette cessation that may ultimately produce an enormous public health impact. We believe the substantial potential benefits significantly outweigh the minimal potential risks to research participants.

# Payment for participation

There is no payment for study enrollment or completion of the baseline assessment. All participants in both arms are asked to complete follow-up surveys at 1- month and 7-months post-randomization. Participants will be paid \$20 for completing each follow-up survey via the Internet or over the phone with a telephone interviewer. Participants who respond within 24 hours of receiving the initial survey invitation will receive an additional \$10. All participants in both arms will also be compensated \$5 for each text message assessment (7 total) they respond to, for a total compensation of up to \$95 for their entire study participation.

Payment for completing the surveys will be delivered via Rybbon, a company specializing in digital gift management for marketing and research. Rybbon is fully integrated with Qualtrics. When a participant completes a follow-up survey via Qualtrics, Rybbon will generate a unique link for giftcard redemption and will email it to the participant. Rybbon has no access to any other identifying

information other than email and no access to survey data. Participants can redeem their Rybbon giftcard from a variety of giftcard options. Those completing text message assessments will receive a link to a Rybbon payment via text message upon responding to each assessment.

#### IMPORTANCE OF THE KNOWLEDGE TO BE GAINED

This is Quitting is the first text message intervention for e-cigarette cessation designed specifically for young people. We have seen a high volume of enrollment since the program launched in January 2019 with only earned media and organic marketing efforts to date. We have been flooded with interest from youth-serving organizations looking for a proven quit vaping program to offer to their young people. To our knowledge, this study will be the first to rigorously evaluate a scalable, cost-efficient, market-tested quit vaping program among users aged 18-24. These data are urgently needed.

#### DATA AND SAFETY MONITORING PLAN

Confidentiality will be protected at all times and potential risks will be minimized systematically.

## **Data Safety**

Respondents will fill out computer-based surveys. All data collected via surveys will be stored in a secure Qualtrics database online (see **Appendices A & B** for information on data security and storage). All research studies and their related non-public materials are confidential information. This includes, but is not limited to, the study title, study questions that are responded to, provided as part of a study, and any concepts related to those materials. Respondent information will remain confidential.

All data used specifically for this project will be maintained in a manner consistent with NIH standards. The Principal Investigator (Dr. Amanda Graham), Data Analyst (Dr. Michael Amato), Project Managers (Sarah Cha, Megan Jacobs), research assistants (Mia Bottcher, Jenna Woodward), and software development team will have access to participants' identifying information. All study staff will have received certification in human subjects protection from the NIH Office of Human Subjects Research. Confidentiality of data will be maintained by numerically coding all data, by disguising identifying information, and by keeping all data electronically protected. Electronic data files with identifiable information will be maintained separately from other data files and will only be used for administrative purposes. Identifying information will not be reported. The list of participant phone numbers, content of text message responses, and documentation of incoming and outgoing messages will be accessible to study staff through a password protected administrative web page available only over an encrypted connection (SSL).

## **Adverse Event Reporting**

HHS definition for "adverse events" will be used for this study (<a href="https://www.hhs.gov/ohrp/regulations-and-policy/guidance/reviewing-unanticipated-problems/index.html#AA">https://www.hhs.gov/ohrp/regulations-and-policy/guidance/reviewing-unanticipated-problems/index.html#AA</a>). Adverse event is defined as any untoward or unfavorable medical occurrence in a participant, including any abnormal sign, symptom, or disease temporally associated with participation in the research. A serious adverse event is defined as any adverse event temporally associated with the subject's participation in research that: 1) results in death; 2) is life-threatening; 3) requires inpatient hospitalization or prolongation of existing hospitalization; 4) results in a persistent or significant disability/incapacity; 5) results in congenital anomaly/birth defect; or 6) any other adverse event that may jeopardize the participant's health and may require medical or surgical intervention to prevent one of the other outcomes listed above. Unanticipated problem includes any incident, experience, or outcomes that is: 1) unexpected given the research procedures and the characteristics of the subject population being studied; 2) related or possibly related to a subject's participation in the research; and 3) suggest that research places subjects or others at a greater risk of harm related to the research than was previously known or recognized.

Adverse events, serious adverse events, and unanticipated problems are unlikely in this sociobehavioral only intervention, but any potential events will be reported immediately upon discovery by study staff to the Principal Investigator who will notify the IRB within 24 hours.

#### **Regulatory and Ethical Considerations**

This study targets health topic that is currently receiving significant media and regulatory attention (e-cigarette use). We do not anticipate any regulatory changes that may occur during the study period to impact study conduct as our study is aimed at

evaluating a cessation program for a product that may become less available and fits well into the currently developing regulatory environment.

The assessment-only arm was selected as the most ethical control group for the current study that allows for evaluation of the intervention while keeping control arm participants engaged. All control arm participants will have access to the program at the conclusion of the study if they are interested.

Our payment structure was developed to incentivize participants for their time and increase retention while not creating any coercion. Thus the incentives are nominal amounts, but provides choices for participants that we hypothesize will lead to great retention.

The current study is as a low risk, sociobehavioral only intervention and we do not anticipate any other ethical considerations.

#### **RECRUITMENT MATERIALS**

#### **Sample Recruitment Advertisement Text Options**

- Do you JUUL? Interested in quitting? You may be eligible for a paid study! Click here for more info.
- Do you vape? Thinking about quitting? You may be eligible for a paid study. Click here for more info.
- If you've been thinking about quitting JUUL (or whatever vape you used to love), you may be eligible for a paid study. Click to learn more!

### **Study Information Page Text**

We are evaluating a new quit vaping/JUULing program developed by Truth Initiative, America's largest nonprofit public health organization dedicated to making tobacco use a thing of the past. We need your help to make it the best it can be!

#### What would I be asked to do?

- 1. Answer a few questions today to see if you're eligible
- 2. Complete an 8-10 minute survey today about your experience vaping
- 3. Sign up for a text message program and respond to the first message
- 4. Answer a few text message questions over the next 6 months about your vaping/JUULing
- 5. Complete 2 surveys, 1month and 7 months from now to tell us about your vaping/JUULing

## Why should I join the study?

Your feedback will be invaluable in helping us evaluate our program.

To thank you, you'll receive \$5 each time you tell us about your vaping status via text message, and \$30 when you complete the 1-month and 7-month surveys. That's a **total possible \$95**.

This program may also help you in your own efforts to quit vaping/JUULing!

#### How will my information be used?

Your name and the fact that you were in the study will be kept completely confidential. Results of this research study will be used to improve the program. They will also be published in scientific reports and shared at academic conferences.

Ready to answer a few questions to see if you are eligible?

\*\*\*\* CHECK MY ELIGIBILITY \*\*\*\*

WHO WE ARE ▼

WHAT WE DO ▼

OUR TOP ISSUES ▼

RESEARCH & RESOURCES ▼

GET INVOLVED ▼

SEARCH Q

Study

Quit Vaping Study

Nov. 06, 2019

We are evaluating a new quit vaping/JUULing program developed by Truth Initiative, America's largest nonprofit public health organization dedicated to making tobacco use a thing of the past. We need your help to make it the heat it can be for

#### RESEARCH AND EVALUATION

Learn more about that Truth Initiative Schroeder Institute®



#### What would I be asked to do?

- 1. Answer a few questions today to see if you're eligible
- 2. Complete an 8-10 minute survey today about your experience vaping
- ${\bf 3.}\,$  Sign up for a text message program and respond to the first message
- $\textbf{4.} \ \, \text{Answer a few text message questions over the next 6 months about your vaping/JUULing}$
- 5. Complete 2 surveys, 1 month and 7 months from now, to tell us about your vaping/JUULing

# Why should I join the study?

Your feedback will be invaluable in helping us evaluate our program.

To thank you, you'll receive \$5 each time you tell us about your vaping status via text message, and \$30 when you complete the 1-month and 7-month surveys. That's a **total possible \$95**.

This program may also help you in your own efforts to quit vaping/JUULing!

#### How will my information be used?

Your name and the fact that you were in the study will be kept completely confidential. Results of this research study will be used to improve the program. They will also be published in scientific reports and shared at academic conferences.

Ready to answer a few questions to see if you are eligible?

CHECK MY ELIGIBILITY →



# **ASSESSMENTS**

# **Screening Questionnaire**

\* Bolded response options required for eligibility

1. How old are you? (18-24 required for eligibility)

\*\*Please note that the terms "vape" or "vaping" in this survey refer to use of all vaping products, including JUUL, mods, and other ecigarettes.\*\*

| | [numeric entry] |
|---|---|
| 2. | How often do you vape <u>nicotine</u> ? |
| | 1 = Daily or almost daily |
| | 2 = Less than daily, but at least once a week |
| | 3 = Less than weekly, but at least once a month |
| | 4 = Less than monthly |
| | 5 = Not at all |
| | 6 = Don't know |
| 3. | How often do you vape marijuana, marijuana concentrate, marijuana waxes, THC, CBD or hash oil? |
| | 1 = Daily or almost daily |
| | 2 = Less than daily, but at least once a week |
| | 3 = Less than weekly, but at least once a month |
| | 4 = Less than monthly |
| | 5 = Not at all |
| | 6 = Don't know |
| 4. | Are you seriously thinking about quitting vaping? |
| | 1 = Yes, during the next 30 days |
| | 2 = Yes, in the next 6 months |
| | 3 = Yes, in the next 12 months |
| | 4 = Yes, but not in the next 12 months |
| | 5 = No, I'm not thinking about quitting vaping |
| 5. | What is the highest level of school/degree you have completed? |
| | 1 = Less than high school (no diploma) |
| | 2 = GED or equivalent |
| | 3 = High school graduate |
| | 4 = Some college or technical school |
| | 5 = College graduate |
| | 6 = Graduate degree |
| | 7 = Prefer not to say |
| 6. | Considering your income and income from any people who help you, what is your personal financial situation? |
| | 1 = Live comfortably |
| | 2 = Meet needs with a little left |
| | 3 = Just meet basic expenses |
| | 4 = Don't meet basic expenses |
| 7. | What is your gender identity? |
| | 1 = Male |
| | 2 = Female |
| | 3 = Non-binary |
| | 4 = Other 5 = Prefer not to say |
| | 5 = Prefer not to SaV |

| | 1 = Black or African American |
|---|---|
| | 2 = American Indian or Alaska Native |
| | 3 = Asian |
| | 4 = Native Hawaiian/Other Pacific Islander |
| | 5 = White |
| | 6 = Other |
| | 7 = Prefer not to say |
| 9. | Are you Hispanic, Latino/a, or Spanish origin? |
| | 0 = No |
| | 1 = Yes |
| | 2 = Prefer not to say |
| 10 | Which of the following best describes you? |
| 10. | 1 = Straight |
| | 2 = Gay or lesbian |
| | 3 = Bisexual |
| | 4 = Other |
| | 5 = Prefer not to say |
| | 5 - Therefi flot to say |
| Thanks | following message. for your interest in the study but unfortunately you are not eligible. For free help quitting vaping, text DITCHJUUL to 88709. |
| **** | |
| Participo | ants who are <b>eligible</b> will see the following message and receive a link via email to complete the Baseline Survey. |
| You are | eligible for the study! The next step is a short survey. Please enter your email and we'll send a link to the survey. |
| | Email: |
| | Confirm your email: |
| | the cell phone number where you want to receive our text messages? **Please make sure to use this same phone number when up to enroll in the study** |
| | Cell phone number: |

8. Which of the following would you say is your race? Check all that apply.

#### **Baseline Assessment**

\*\*The terms "vape" or "vaping" in this survey refer to all vaping products, including JUUL, mods, and other e-cigarettes.\*\*

#### ADDITIONAL DEMOGRAPHIC QUESTIONS

- 1. Are you currently a student?
  - 1 = No
  - 2 = Yes
  - 3 = Prefer not to say
- 2. [SKIP PATTERN, Only ask if YES to Q1] What school do you currently attend?
  - 1 = High school
  - 2 = Vocational/technical school
  - 3 = Community college or junior college
  - 4 = 4-year college or university
  - 5 = Graduate or professional school
  - 6 = Other (specify):
  - 7 = Prefer not to say
- 3. Which best describes your current job/paid employment status?
  - 1 = Work full-time (35 hrs/wk or more)
  - 2 = Work part-time (15-34 hrs/wk)
  - 3 = Work part-time (less than 15 hrs/wk)
  - 4 = Don't currently work for pay
  - 5 = Prefer not to say

#### **E-CIGARETTE USE HISTORY**

#### These questions are all about vaping NICOTINE.

- 4. How many days per week do you vape? [Integer response, 1-7]
- 5. On average, how many puffs/hits on your vape do you take on a typical day? [Integer response, any]
- 6. On average, how much do you spend a week on vaping? \$[integer response, any]

## **CONFIDENCE/MOTIVATION/SELF-EFFICACY**

- 7. How much do you want to quit vaping?
  - 1 = Not at all
  - 10 = Very much
- 8. How confident are you that you can quit vaping?
  - 1 = Not at all
  - 10 = Very much
- 9. Which of these statements apply to you? Select all that apply.
  - 1 = I vape to cope with stress
  - 2 = I am scared about quitting vaping
  - 3 = Sometimes I think quitting vaping will be impossible
  - 4 = I want to quit vaping but I don't know how

# **PAST QUIT ATTEMPTS**

These questions are all about vaping NICOTINE.

- 10. In the past 12 months, how many times have you stopped vaping for one day or longer?
  - 1 = None
  - 2 = 1 time
  - 3 = 2 times
  - 4 = 3 to 5 times
  - 5 = 6 to 9 times
  - 6 = 10 or more times
- 11. In the past 12 months, has a doctor/dentist/etc advised you to quit vaping?
  - 0 = No
  - 1 = Yes
  - 2 = I haven't seen a doctor/dentist/etc in the past 12 months
- 12. How much do you want to quit vaping because...

| men men de jeu mant te dant raping secondesin | |
|---|---|
| It's bad for your health. | 1 = Not at all, 10 = Very much |
| It's too expensive. | 1 = Not at all, 10 = Very much |
| It's difficult to get (e.g. device, e-liquid, pods, | 1 = Not at all, 10 = Very much |
| cartridges) | |
| Someone else is making me quit | 1 = Not at all, 10 = Very much |
| I want to quit for someone else. | 1 = Not at all, 10 = Very much |
| I don't want to be punished for vaping | 1 = Not at all, 10 = Very much |
| I don't want to be addicted. | 1 = Not at all, 10 = Very much |
| It's just wrong for me to use it. | 1 = Not at all, 10 = Very much |
| Other: | 1 = Not at all, 10 = Very much |

# **E-CIGARETTE DEPENDENCE**

| | Never | Rarely | Sometimes | Often | Almost always |
|---|---|---|---|---|---|
| 13. I find myself reaching for my vape without thinking about it. | 0 | 1 | 2 | 3 | 4 |
| 14. I drop everything to go out and buy a vape or e-liquid | 0 | 1 | 2 | 3 | 4 |
| 15. I vape more before going into a situation where vaping is not allowed. | 0 | 1 | 2 | 3 | 4 |
| 16. When I haven't been able to vape for a few hours, the craving gets intolerable. | 0 | 1 | 2 | 3 | 4 |

| 17. Have you ever tried to stop vaping, but couldn't? | Yes | No |
|---|---|---|
| 18. Do you vape now because it is really hard to quit? | | |
| 19. Have you ever felt like you were addicted to vaping? | | |
| 20. Do you ever have strong cravings to vape? | | |
| 21. Have you ever felt like you really needed to vape? | | |
| 22. Is it hard to keep from vaping in places where you are not supposed to, like school or work? | | |
| When you tried to stop vaping (or when you haven't vaped in awhile) | | |
| 23. Did you find it hard to concentrate because you couldn't vape? | | |
| 24. Did you feel more irritable because you couldn't vape? | | |
| 25. Did you feel a strong need or urge to vape? | | |
| 26. Did you feel nervous, restless or anxious because you couldn't vape? | | |

| 27. | How soon as you wake up do you first vape? 1 = Within 5 minutes 2 = 6 to 30 minutes 3 = 31 to 60 minutes 4 = After 60 minutes |
|---|---|
| 28. | How aware are you of media reports on illnesses and deaths related to vaping? 1 = Not at all 10 = Very much |
| 29. | How worried are you about the consequences of vaping? 1 = Not at all 10 = Very much |
| 30. | Have you experienced any of the following vaping-related symptoms? Select all that apply. 1 = Respiratory symptoms (e.g., cough, chest pain, and shortness of breath) 2 = Gastrointestinal symptoms (e.g., abdominal pain, nausea, vomiting, and diarrhea) 3 = Fever, chills, or weight loss |
| soc | CIAL SUPPORT |
| 31. | Of the 5 closest friends you spend time with on a regular basis, how many of them vape NICOTINE? [Dropdown 1-5] |
| 32. | Does anyone who lives with you vape NICOTINE? 1 = Yes 2 = No |
| 33. | Does anyone who lives with you now use other tobacco products, like cigarettes, cigars, chewing tobacco, etc?<br>1 = Yes<br>2 = No |
| 34. | How many of your <u>friends</u> are supportive of your desire to quit vaping? 1 = All of them 2 = Most of them 3 = About half of them 4 = Very few of them 5 = None of them 6 = No one knows I want to qui |
| 35. | How many of your <u>family members</u> are supportive of your desire to quit vaping? 1 = All of them 2 = Most of them 3 = About half of them 4 = Very few of them 5 = None of them 6 = No one knows I want to quit |
| 36. | Which of the following statements apply to you? Select all that apply. 1 = I feel pressured to vape from my friends 2 = I have been teased/bullied for wanting to quit 3 = Most people my age who vape don't want to quit 4 = Thinking about quitting makes me feel alone |
| 37. | Out of 100 people your age, how many of them do you think vape? |

1 = Nearly all of them 2 = Most of them

- 3 = About half of them
- 4 = Less than half of them
- 5 = Almost none of them
- 38. Out of 100 people your age who vape, how many of them do you think want to quit?
  - 1 = Nearly all of them
  - 2 = Most of them
  - 3 = About half of them
  - 4 = Less than half of them
  - 5 = Almost none of them

#### **OTHER SUBSTANCE USE**

39. During the past 30-days (including today), did you use any of these products, even once?

| | No | Yes |
|---|---|---|
| Large cigars (like Cohiba or Romeo y Julieta) | 0 | 1 |
| Little cigars/cigarillos (e.g., Black and Milds, Swisher Sweets, Dutch Masters, Phillies Blunts) | 0 | 1 |
| Cigarettes | 0 | 1 |
| Hookah/shisha/waterpipe (hookah tobacco) | 0 | 1 |
| Chewing tobacco, snuff, or snus | 0 | 1 |
| Marijuana/cannabis | 0 | 1 |

- 40. Have you ever, even once, had a drink of any type of alcoholic beverage? Please do not include times when you only had a sip or two from a drink.
  - 1 = Yes
  - 2 = No
- 41. How long has it been since you last drank an alcoholic beverage?
  - 1 = Within the past 30 days
  - 2 = More than 30 days but within the past 12 months
  - 3 = More than 12 months ago
- 42. What's your best estimate of the # of days you drank alcohol during the past 30 days?
  - 1 = 1 or 2 days
  - 2 = 3 to 5 days
  - 3 = 6 to 9 days
  - 4 = 10 to 19 days
  - 5 = 20 to 29 days
  - 6 = All 30 days
- 43. On the days you drank in the past 30 days, how many drinks did you usually have each day?



drinks

| 44. | In the past 30 days, | on how many days did | you have 4 (fe | males)/5 (males) ( | or more drinks on | the same of | occasion? |
|---|---|---|---|---|---|---|---|
| | days | | | | | | |

# **MENTAL HEALTH CO-MORBIDITIES**

45. In the last 2 weeks, how often have you been bothered by any of the following?

| | Not at all | Several days | More than half the days | Nearly every<br>day |
|---|---|---|---|---|
| Little interest or pleasure in doing things | 0 | 1 | 2 | 3 |
| Feeling down, depressed, or hopeless | 0 | 1 | 2 | 3 |
| Feeling nervous, anxious or on edge | 0 | 1 | 2 | 3 |
| Not being able to stop or control worrying | 0 | 1 | 2 | 3 |

- 46. What's your MAIN reason for joining this research study?
  - 1 = I want to learn more about vaping
  - 2 = I want to quit vaping
  - 3 = I want to make money
  - 4 = I'm interested in research

#### **Follow-Up Assessment**

\* Only items not repeated from Baseline Assessment are noted below

#### **ABSTINENCE STATUS AND MOTIVATION TO QUIT**

\*\*Please note that the terms 'vape' or 'vaping' in this survey refer to use of all vaping products, including JUUL, mods, and other ecigarettes.\*\*

For these questions, please think of your use of vape that contain nicotine only in your responses. OK, let's get started!

- 1. In the past 30 days, did you vape at all, even a puff of someone else's?
  - 0 = No
  - 1 = Yes
- 2. [Skip logic, only ask if Q1 = Yes] Have you used any vape, even one puff, in the past 7 days?
  - 0 = No
  - 1 = Yes
- [Skip logic, only ask if Q1 or Q2 = No] When was the last time you vaped?[Enter date]

## **QUIT METHODS**

- 4. [Since you joined the study a month ago/In the last 6 months], how many times have you stopped vaping not even a puff for one day 24 hours or longer because you were trying to quit for good?
  - \*\*Please note! We're looking for the **number of quit attempts** you've made, not the number of days you've been quit. For example, if you quit once and stayed quit for a week, please enter 1 (not 7).\*\*
  - quit attempt(s) [numeric entry]
- 5. [Skip logic, only ask if response to Q4 > 0] In the past [1/6 months], which of the following things have you tried to quit vaping? Check all the categories that apply.
  - Nicotine replacement medicine (patch, gum, lozenge, nasal spray, inhaler)
  - Prescription medicine like Zyban/bupropion or Varenicline/Chantix
  - Switching to cigarettes
  - Switching to chewing tobacco or snuff
  - Quit vaping text message program NOT part of this study
  - Other (specify):
  - None of the above

#### **CUSTOMER SATISFACTION QUESTIONS**

- 6. Overall, how satisfied are you with the guidance and information you received from the quit vaping text message program?
  - 1 = Very satisfied
  - 2 = Somewhat satisfied
  - 3 = A little satisfied
  - 4 = Not at all satisfied
- 7. How likely would you be to recommend the quit vaping text message program to family or friends who want to quit JUULing/vaping?? 0-10 scale
- 8. Was the number of text messages from the quit vaping text message program too many, too few, or just right?
  - 1 = Too few
  - 2 = Just right
  - 3 = Too many

9. Based on your experience with the text messages from This is Quitting, how much do you agree/disagree with the statements below?

| | Completely | Agree | Disagree | Completely |
|---|---|---|---|---|
| | agree | somewhat | somewhat | disagree |
| | (4) | (3) | (2) | (1) |
| They helped me stay on track with quitting | | | | |
| They helped me feel more confident about | | | | |
| quitting | | | | |
| They were written personally for me | | | | |
| They suggested quitting strategies that were new | | | | |
| to me | | | | |
| They made me feel less alone in quitting | | | | |
| They made me feel that I knew the right steps to | | | | |
| take to quit | | | | |
| I liked being able to interact with the text | | | | |
| messages | | | | |
| I liked reading tips from other people who had | | | | |
| quit | | | | |

## **BRAND AWARENESS**



10. Do you recognize this logo?

0 = No

1 = Yes

11. [If YES to #10] What do you think of when you see this logo? Select all that apply.

- 1 = Anti-alcohol
- 2 = Anti-drunk driving
- 3 = Anti-drug
- 4 = Anti-tobacco
- 5 = Anti-vape
- 6 = Anti-e-cigarettes (including JUUL)
- 7 = None of these [EXCLUSIVE]
- 8 = Not sure [EXCLUSIVE]

12. [If YES to #10] How much do you agree or disagree with the following? 1 = Strongly disagree, 3 = Neither agree/Disagree, 5 = Strongly agree

- I'd like to help truth make a difference in my generation
- I'd defend truth on social media if someone were putting it down
- I'd follow truth on social media
- I would be part of a movement that embraces informed decision making
- Truth is helping my generation make informed choices
- Truth is for people like me



| 13. | Do you recognize this logo? 0 = No 1 = Yes |
|---|---|
| | 1 - 163 |
| 14. | [If YES to #13] What do you think of when you see this logo? Select all that apply. 1 = Anti-alcohol 2 = Anti-drunk driving 3 = Anti-drug 4 = Anti-tobacco 5 = Anti-vape 6 = Anti-e-cigarettes (including JUUL) 7 = None of these [EXCLUSIVE] 8 = Not sure [EXCLUSIVE] |
| 15. | [If YES to #13] To your best knowledge, what is <b>This is Quitting</b> ? Select all that apply. |
| | 1 = A website |
| | 2 = A text message program |
| | 3 = A class you can take through school |
| | 4 = A mobile app 5 = No clue [EXCLUSIVE] |
| 16. | Are you familiar with the hashtags #ditchjuul, #ditchvape, or #ThisisQuitting? |
| | 0 = No |
| | 1 = Yes |
| 17. | Have you used any quit vaping text message program other than what you received for this research study? 0 = No 1 = Yes |
| 18. | [If YES to #17] What was the text message program you used? [open ended short entry] |
| <u>CO\</u> | /ID-19 RELATED ITEMS? |
| The | next few questions are related to other health issues that may be related to vaping/quitting vaping. |
| 19. | Please use the following scale to indicate your current thoughts about vaping and COVID-19. 0 = Not at all to 10 = Extremely |
| | How concerned about COVID-19 are you for your own health? |
| | How concerned about COVID-19 are you for others' health? |
| | • How much do you believe your vaping (now or in the past) increases your risk of harm from COVID-19? |
| 20. | Has any of the following changed since learning about COVID-19? 1 = Decreased, 2 = Remained the same, 3 = Increased • My motivation to quit • My use of vape • My access to vape |
| 21. | How has the COVID-19 pandemic made it easier or harder to quit vaping? [open ended text entry] |

| 22. | Awesome, you're done! Any other feed | , _ | We're always looking to improve | e, so your ideas are welcome. |
|---|---|---|---|---|
| <u>REIV</u> | MINDER MESSAGE RE: PAYMENT | | | |

Thanks again for your time and feedback. Click the following link to select the incentives that you want to receive. If you completed your survey within 24 hours of receiving the notice, we will send you a separate note to about your extra \$10 bonus. If you have any questions, please send us a note at <a href="mailto:vapestudy@truthinitiative.org">vapestudy@truthinitiative.org</a>.

Thanks!

~ Sarah (Research Manager for the Truth Initiative Quit Vaping Study)

\*\*LINK TO RYBBON\*\*

# **EXIT QUESTIONNAIRE POST 7-MONTH ASSESSMENT ONLY**

1. How important was each of these reasons for joining the study?

| | | 0 = Not<br>important<br>at all | 1 | 2 | 3 = Very<br>important |
|---|---|---|---|---|---|
| The money | | | | | |
| Soi | unded interesting | | | | |
| Wa | Wanted to cut down/quit vaping | | | | |
| Liked Truth Initiative/This is Quitting | | | | | |
| Someone I know wanted me to join | | | | | |
| | | | | | _ |
| 2. | How closely did you pay attention to the study questions and your answers? | 1 = I did not<br>pay<br>attention | 2 | 3 | 4 = I paid<br>close<br>attention |
| | | | | | <del>,</del> |
| 3. | How much do you like or dislike the way vaping makes you look? | 1 = Dislike<br>very much | 2 | 3 | 4 = Like very<br>much |
| | | | | | _ |
| 4. | Did you have any concerns about confidentiality in the study, i.e. whether information you provided would be shared with parents or others? | 1 = Not<br>concerned<br>at all | 2 | 3 | 4 = Very<br>concerned |
| | | | | | <del> </del> |
| 5. | How important was it for the study team to like you? | 1 = Not<br>important<br>at all | 2 | 3 | 4 = Very<br>important |

- 6. Did you ever feel the study team wanted you to report that you vaped...
  - 1 = Less than you actually did
  - 2 = As much as you actually did
  - 3 = More than you actually did

# **SAMPLE TEXT MESSAGES**

| Message type | Sample messages |
|---|---|
| No quit date | |
| Building skills | For one day, keep track of when you [device] and what the situations are that make you crave or [device]. By knowing your triggers, you can make plans to deal with those *without* your [device]. |
| Confidence | Anon says "You are strong, you deserve freedom from addiction. And it's time for us to own that." You CAN do this. Maybe right now isn't the right time for you to quit, but stick with me for a few more weeks I'll send tips to help you feel more ready. |
| Has quit date | |
| Encourage and support | Benji says "If I can quit anyone can quit there's no way anyone is ever been as addicted as I was." No matter how much you use an [device], it's definitely possible to quit. |
| Skill- and self-efficacy building exercises | AnnetteMM says "Gather preparation supplies ahead of time. I bought twizzlers and tootsie pops." Tell me what you're going to buy to put in your mouth instead of a [device] next week. |
| Coping strategies | If you used to [device] a lot, you might feel anxious or sweaty today. Keep taking deep breaths and drinking cold water. It's going to be ok you can get through today. |
| Information about risks of vaping | Pam loves to walk and hike, and her [device] felt like it got her heart racing or she felt nervous. Quitting will help you feel like the best version of you. |
| Benefits of quitting | Brittany suggests keeping track of how much money you used to spend on your [device] so you can see what you're saving. Makes you feel rich! |
| Cutting down to quit | SpartanGirl117 says "It takes time to break the habit so be patient. Each time you beat a craving, your brain is relearning a new habit of NOT using your [device]" |
| On-demand support | |
| COPE | tjh.upnext says "I like to keep a water on me. End one addiction with another one. Drink water when you are having an urge. Healthy addiction!" |
| STRESS | Chase says "It's alright take it a few minutes at a time if you are stressed remember it only last a few minutes at a time" |
| SLIP | Practice makes progress! This is a process, and you're still learning what the right way is for YOU to quit. |
| MORE | • jklause says "Remember why your quitting and don't look back. Keep going |
| • FEELS | strong and you'll be able to achieve sobriety." |
| • TIPS | <ul> <li>Anonymous says "Make a list of reasons as to why you want to quit. Have it<br/>on your phone or carry it around, and read over it during a craving."</li> </ul> |

#### PARTICIPANT COMMUNICATION

#### **Confirmation Email with Link to Baseline**

Subject: We want you in the Truth Initiative Quit Vaping Study!

Dear {{ participant.name }},

We want you to participate in the Truth Initiative Quit Vaping Study! Your participation will help us build the best quit vaping program possible.

Please fill out the baseline survey by clicking on the link below. You must complete the survey within <u>24 hours</u> to fully enroll in the study!

{{ survey\_link }}

On behalf of the Truth Initiative Quit Vaping Study team, thank you!

Sarah Cha

Project Manager | Truth Initiative Quit Vaping Study | (202) 525-6473

P.S. If for any reason your survey session expires before completing the survey, your answers will be saved and you can finish the survey by clicking on this link again.

## **Survey Invitations**

### Email 1

Subject: It's Sarah from the Truth Initiative Quit Vaping Study – Your survey is waiting!

Dear {{ name }},

It's Sarah from the Truth Initiative Quit Vaping Study - thanks for being a part of our research! It's time for your follow-up survey. It will only take around 10 minutes.

Click or copy/paste the following link to access your unique survey: {{ followup\_url }}

To thank you for your time, we will email you a \$20 gift code to use at an online retailer of your choice. BONUS! We'll add an extra \$10 bonus if you complete the survey within the <u>next 24 hours!</u>

We're evaluating this program, not you. So if you're still vaping or haven't totally quit yet, we still value your response.

Sincerely,

Sarah Cha

Project Manager | Truth Initiative Quit Vaping Study | (202) 525-6473

#### Email 2

Subject: Your response matters! Take the Truth Initiative Quit Vaping Study survey

Dear {{ name }},

Just a quick reminder to complete the follow-up survey for the Truth Initiative Quit Vaping Study. It takes less than 10 minutes to complete and I'll send you a \$20 online gift card (think Amazon, Apple, Target, Starbucks... your choice!).

Click or copy/paste the following link to access your unique survey: {{ followup\_url }}

Thanks so much,

Sarah Cha

Project Manager | Truth Initiative Quit Vaping Study | (202) 525-6473

P.S. Even if you haven't quit vaping, that's OK! Your responses still really matter to our study.

#### Email 3

Subject: \$20 to complete the Truth Initiative Quit Vaping Survey

Dear {{ name }},

I promise: no more emails after this. Please take 10 minutes to fill out the follow-up survey for the Truth Initiative Quit Vaping Study. I'll send you a \$20 gift card to the retailer of your choice.

Click or copy/paste the following link to access your unique survey: {{ followup\_url }}

Your responses are truly valuable to our research, that will help thousands of other young vapers quit. Thank you!

#### Sarah Cha

Project Manager | Truth Initiative Quit Vaping Study | (202) 525-6473

P.S. Not sure if you should take the survey because you haven't quit or are vaping sometimes? Easy answer: YES! Your responses mean so much to our research.

## **Text Message Assessments**

| Time | Original message | Response to anyone sending a response |
|---|---|---|
| 2 weeks Checking in: Have you cut down how much you vape | | Thanks for your time in responding, it's really helpful |
| | nicotine in the past 2 weeks? Respond w/letter: A=I | for our study! We'll be sending you a link to redeem |
| | still use the same amount, B=I use less, C=I don't use | your \$5 incentive shortly. |
| | at all anymore | |
| 1 month – 6 months | How's the quit going? When was the last time you | Thanks for your time in responding, it's really helpful |
| | vaped nicotine, even a puff of someone else's? | for our study! We'll be sending you a link to redeem |
| | Respond w/ letter: A- in the past 7 days, B- 8-30 days | your \$5 incentive shortly. |
| | ago, C- More than 30 days ago | |

#### **REFERENCES**

- 1. Surgeon General's Advisory on E-cigarette Use Among Youth. 2018. at <a href="https://e-cigarettes.surgeongeneral.gov/documents/surgeon-generals-advisory-on-e-cigarette-use-among-youth-2018.pdf">https://e-cigarettes.surgeongeneral.gov/documents/surgeon-generals-advisory-on-e-cigarette-use-among-youth-2018.pdf</a>.)
- 2. Centers for Disease Control and Prevention. Electronic cigarettes: What's the bottom line? 2019.
- 3. Vallone DM, Bennett M, Xiao H, Pitzer L, Hair EC. Prevalence and correlates of JUUL use among a national sample of youth and young adults. Tobacco control 2018.
- 4. In: Eaton DL, Kwan LY, Stratton K, eds. Public Health Consequences of E-Cigarettes. Washington (DC)2018.
- 5. Primack BA, Shensa A, Sidani JE, et al. Initiation of Traditional Cigarette Smoking after Electronic Cigarette Use Among Tobacco-Naive US Young Adults. Am J Med 2018;131:443 e1- e9.
- 6. Gray KM, Baker NL, McClure EA, et al. Efficacy and Safety of Varenicline for Adolescent Smoking Cessation: A Randomized Clinical Trial. JAMA Pediatr 2019.
- 7. Fanshawe TR, Halliwell W, Lindson N, Aveyard P, Livingstone-Banks J, Hartmann-Boyce J. Tobacco cessation interventions for young people. Cochrane Database Syst Rev 2017;11:CD003289.
- 8. Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y, Dobson R. Mobile phone text messaging and app-based interventions for smoking cessation. Cochrane Database Syst Rev 2019;10:CD006611.
- 9. Graham AL, Jacobs MA, Amato MS. Engagement and 3-month outcomes from a digital e-cigarette cessation program in a cohort of 27,000 teens and young adults. Nicotine & tobacco research: official journal of the Society for Research on Nicotine and Tobacco 2019.
- 10. Mendel J. Finding truth in smoking status self-reporting: A formative evaluation of reporting modality used in the Be Free Smoking Study of the Text2Quit program: School of Public Health and Health Services, The George Washington University; 2013.
- 11. Graham AL, Papandonatos GD. Reliability of internet- versus telephone-administered questionnaires in a diverse sample of smokers. Journal of medical Internet research 2008;10:e8.
- 12. Graham AL, Papandonatos GD, Bock BC, et al. Internet- vs. telephone-administered questionnaires in a randomized trial of smoking cessation. Nicotine & tobacco research: official journal of the Society for Research on Nicotine and Tobacco 2006;8 Suppl 1:S49-57.
- 13. Pearson JL, Hitchman SC, Brose LS, et al. Recommended core items to assess e-cigarette use in population-based surveys. Tobacco control 2018;27:341-6.
- 14. Bold KW, Sussman S, O'Malley SS, et al. Measuring E-cigarette dependence: Initial guidance. Addictive behaviors 2018;79:213-8.
- 15. Centers for Disease Control and Prevention. National Youth Tobacco Survey Questionnaire. 2018.
- 16. Morean M, Krishnan-Sarin S, O'Malley SS. Comparing cigarette and e-cigarette dependence and predicting frequency of smoking and e-cigarette use in dual-users of cigarettes and e-cigarettes. Addictive behaviors 2018:87:92-6.
- 17. Case KR, Mantey DS, Creamer MR, Harrell MB, Kelder SH, Perry CL. E-cigarette- specific symptoms of nicotine dependence among Texas adolescents. Addictive behaviors 2018;84:57-61.
- 18. Substance Abuse and Mental Health Services Administration. National Survey on Drug Use and Health Questionnaire. 2018.
- 19. National Health Interview Survey. 2015. (Accessed 06/23/2015, 2015, at http://www.cdc.gov/nchs/nhis/nhis/questionnaires.htm.)
- 20. Abroms LC, Boal AL, Simmens SJ, Mendel JA, Windsor RA. A Randomized Trial of Text2Quit: A Text Messaging Program for Smoking Cessation. American journal of preventive medicine 2014.
- 21. Strecher VJ, McClure J, Alexander G, et al. The role of engagement in a tailored web-based smoking cessation program: randomized controlled trial. Journal of medical Internet research 2008;10:e36.
- 22. Dijkstra A, Ballast K. Personalization and perceived personal relevance in computer-tailored persuasion in smoking cessation. British journal of health psychology 2012;17:60-73.
- 23. Lantini R, McGrath AC, Stein LA, Barnett NP, Monti PM, Colby SM. Misreporting in a randomized clinical trial for smoking cessation in adolescents. Addictive behaviors 2015;45:57-62.
- 24. Blankers M, Smit ES, van der Pol P, de Vries H, Hoving C, van Laar M. The Missing=Smoking Assumption: A Fallacy in Internet-Based Smoking Cessation Trials? Nicotine & tobacco research: official journal of the Society for Research on Nicotine and Tobacco 2016;18:25-33.

#### **APPENDIX A**

# **Privacy and Terms of Service**

HERE COMES A LOT OF **LEGAL MUMBO**. SO, EVEN IF YOU'RE BORED TO TEARS, READ IT AND THEN CHECK OUT THE REST OF OUR WEBSITE.

#### **Privacy Policy**

<u>www.thetruth.com</u> is a website of Truth Initiative, which is dedicated to achieving a culture where all youth and young adults reject tobacco. We respect your privacy and have created this Privacy Policy to explain what information we collect through the website and how we use it. If you have any questions about this policy, please <u>contact us</u>.

## Non-Personally Identifiable User Information

We automatically collect non-personally identifiable information about our site's users, including the domain name and IP address of visitors, the browser and operating system used, the date and time of each visit and the source of referral. This information does not identify individual visitors, and it is used for our own research purposes and to improve the site's content, structure, and security.

#### Cookies

Cookies are information files that allow websites to remember users' activities on a website. When you visit our site, we may send one or more cookies to your computer that uniquely identifies your browser. We use the information we learn from cookies to improve the quality of our service, for example, by tracking user trends. We do not use cookies to track user activity on an individual basis. Most browsers are initially set up to accept cookies, but you can reset your browser to refuse all cookies or to indicate when a cookie is being sent. However, some of our features and services may not function properly if your cookies are disabled.

#### Personally Identifiable Information

We collect personally identifiable information from you through the site (such as your name, mailing address or email address) when you choose to sign up for our newsletter or otherwise voluntarily provide such information to us. We use your personally identifiable information to create a customized digital experience through the various truth platforms, for analytics, personalization and tracking, and for the purpose for which it was provided, (for example, to add you to our newsletter distribution list, to respond to a query or to fulfill a purchase of truth merch). If you provide us with your email address, we may begin sending you emails with information that we think will be of interest to you. If, at any time, you wish to stop receiving emails from us, please follow the unsubscribe instructions at the bottom of any email you receive. If you provide your cell phone number to us, you consent to receive autodialed messages and texts at that number on any subject from us, unless and until you request that such messages stop.

We also use personal information about users to our website to better understand how people use our site so that we can improve the website and its offerings.

Unfortunately, given the complexity of privacy regulations outside the United States, we do not profile, personalize, track or create customized digital experience for IP addresses that appear to come from outside the United States. As a result, you may not have the benefit of full digital platform experience.

## Security

We take appropriate security measures to protect against unauthorized access to or disclosure or destruction of our users' data. We restrict access to personal information to our employees, contractors, and agents who need to know that information in order to perform their jobs. Nonetheless, we cannot guarantee that your information is 100% secure.

#### **Sharing Personal Information**

We may share your personal information with other like-minded organizations, government officials or other policy-makers, or the press if we believe it will help advance our mission of achieving a culture where all youth and young adults reject tobacco and drugs.

We may also share your information if you provide the information in a context where you would expect the information to be shared. For instance, if you choose to sign a truth-sponsored petition with your name and email address, we may share that information with the party receiving the petition. We may use third party service providers to help us operate our website or administer activities on our behalf. Examples may include fulfilling orders, delivering packages, removing repetitive information from customer lists, processing credit card payments and providing customer service. We may share personal information about our users with these third parties for those limited purposes, but we require that such third parties protect the confidentiality of user information and use it for no other purpose.

In addition, we will share personally identifiable information about our users when required to do so by law, or in the good faith belief that such action is necessary to comply with state and federal laws or to respond to a court order, subpoena, or search warrant. We will also share personally identifiable information if we believe it is necessary to protect the rights, property and safety of us or others.

We may also share personally identifiable information in connection with, or during negotiations of, a merger, sale of company assets, financing or acquisition of all or a portion of our business to another entity. Moreover, we may share personally identifiable information about a user upon the user's consent.

We may share generic aggregated demographic information not linked to any personally identifiable information regarding our website users with third parties.

## Third Party Websites

We may reference mobile applications ("apps") or provide links from our website to other websites. We do not control the content or links that appear on these third party websites/apps, and we are not responsible for the practices employed by websites linked to or references to apps from our site. For instance, these other websites/apps may use cookies or other methods to track and profile people. These third-party websites and services have their own privacy policies. Browsing and interaction on any other website and/or app, including websites that have a link to or apps referenced from our site, is subject to that website's/app's own terms and policies. This Privacy Policy covers only information collected through the use of this website. In addition, we do not currently respond to web browser "do not track" signals.

## Adobe Cloud Marketing Coop

Truth Initiative participates in the Adobe Marketing Cloud Device Co-op to better understand how you use our website and apps across the various devices you use, and to deliver tailored promotions and communications. Learn more at <a href="https://cross-device-privacy.adobe.com">https://cross-device-privacy.adobe.com</a> about how Adobe does this.

## Compliance with Children's Online Privacy Protection Act

Protecting the privacy of the young is especially important. For that reason, we never collect information at the website from those we know are under 13, and no part of the website is structured to attract anyone under 13. If we become aware of having information about anyone under 13, we will promptly delete the information, unless we obtain consent from the parent or legal guardian of the child to retain such information.

#### SPECIAL PROVISIONS FOR THIS IS QUITTING PROGRAM

We are excited that you have decided to use This is Quitting to achieve your vaping cessation goals. We are constantly trying to improve our web and mobile tools to help people quit vaping. To further that goal, we collect data about your use of This is Quitting services (e.g., number and frequency of program use, the content of your texts, etc.).

Data collected from the program may be used for public health and research purposes to help us build better tools for quitting smoking or vaping.

When you sign up for This is Quitting, you are agreeing that at a later date, we may send you communications and content about other Truth Initiative programs, initiatives, campaigns and messaging. You may unsubscribe to these communications at any time.

We may share with other third-party research partners or sponsoring organizations certain aggregated, de-identified data collected from users without their consent. Such information will not include any personally identifiable information such as your name or phone number.

Information provided as part of This is Quitting does not constitute medical advice. This is Quitting services are not to be used to make diagnoses, prescribe medicine or provide treatment, and should not be relied upon as a substitute for consultations with qualified health professionals who are familiar with your individual medical needs. The This is Quitting program is provided as a self-help service to provide you with support while quitting vaping. Please contact your health care provider with any concerns about your physical or mental health or about whether this program is or is not working for you. We do not promise or guarantee any outcome, including that you will successfully quit vaping.

For versions of This is Quitting offered through a school, healthcare system, public health organization or other sponsoring entity (each, a "Sponsoring Entity"), we may share aggregated, de-identified data about your use of This is Quitting with such Sponsoring Entity.

### CHANGES TO THIS PRIVACY POLICY

We may update this Privacy Policy at any time. When we do, we will revise the updated date at the bottom of this page. We encourage our website users to frequently check this page for any changes to stay informed about what information we collect and how we use that information. You acknowledge and agree that it is your responsibility to review this Privacy Policy periodically and become aware of any modifications since your last visit. Your further use of this site following any such modifications constitutes your agreement to the terms of the amended Privacy Policy.

#### Your Acceptance of These Terms

By using this website, you signify your acceptance of this Privacy Policy. If you do not agree to this policy, please do not use the website. Your continued use of the site following the posting of changes to this Privacy Policy will be deemed your acceptance of those changes.

#### **Terms of Service**

Truth Initiative provides the website <u>www.thetruth.com</u> (the "Site") under the following Terms of Service ("Terms"), which may be amended from time to time at our sole discretion. Your use of the Site constitutes your agreement to these Terms.

#### *Intellectual property*

Unless otherwise indicated, Truth Initiative owns all legal right, title and interest in and to the Site, including any and all intellectual property rights. All such intellectual property, including without limitation all trademarks of Truth Initiative, may not be used without Truth Initiative's written consent.

#### User-Provided Content

You, not Truth Initiative, are legally responsible for any material you post on the Site ("Your Content"). You agree to post only content to which you own the copyright (or other applicable rights) or have written permission from the rights owner to post. Your Content also encompasses your name, likeness and/or image, should you post such items to the Site. You agree not to post any material that:

- violates or infringes upon the intellectual property, privacy, publicity or similar rights of others;
- is abusive, offensive, discriminatory, profane, vulgar, obscene, disparaging, defamatory, libelous, slanderous, or contains information known by you to be false, inaccurate, or misleading;
- violates any law, statute, ordinance or regulation or any third party agreement to which you are subject (e.g., Facebook, Twitter, Instagram, Vine, YouTube, Pinterest, etc.);
- contains (i) third party websites; and/or (ii) addresses, email addresses, contact information, phone numbers or other personal identifiable information (other than your own);
- is in the nature of advertising or marketing; and/or
- contains any computer viruses, worms, harmful code, or other potentially damaging computer programs, applications or files.

In addition, by posting Your Content on the Site, you grant Truth Initiative a non-exclusive, perpetual and royalty-free right and license to use, store, display, reproduce, modify, create derivative works, perform, and distribute Your Content in any manner consistent with Truth Initiative's charitable purpose. This means that Your Content will not be treated as confidential and proprietary, and we'll be able to freely use Your Content without attribution or compensation or payment of any kind to you.

Truth Initiative does not endorse or take responsibility for user-provided content. While Truth Initiative does not routinely review user-proved content, Truth Initiative reserves the right, but is not obligated, to remove any information or materials posted on the Site for any or no reason, at its sole discretion.

#### You Represent and Warrant That:

- You are at least thirteen (13) years of age;
- You own or otherwise lawfully possess all rights in and to Your Content; and
- Your Content does not and will not violate these Terms or cause injury to any person or entity.

## **Indemnification and Hold Harmless**

You will indemnify and hold harmless Truth Initiative and its officers, directors, employees, and agents from all claims arising out of or related to: (i) Your Content; and/or (ii) your use of, or your inability to use, the Site or the information contained therein or any other website(s) to which the Site is linked.

#### **Modifications**

Truth Initiative reserves the right to change or terminate any aspect of the Site, including the Site itself and individual user accounts for any or no reason. Truth Initiative also reserves the right to impose limits on certain features of the Site or restrict access to all or parts of the Site without notice or penalty. Additionally, Truth Initiative may revise these Terms from time to time, and the most current version will always be posted on the Site.

## **Limitation of Liability**

TO THE MAXIMUM EXTENT PERMITTED BY LAW, TRUTH INITIATIVE SHALL NOT BE LIABLE FOR ANY INDIRECT, INCIDENTAL, SPECIAL, CONSEQUENTIAL OR PUNITIVE DAMAGES, OR ANY LOSS OF PROFITS OR REVENUES, WHETHER INCURRED DIRECTLY OR INDIRECTLY, OR ANY LOSS OF DATA, USE, GOOD-WILL, OR OTHER INTANGIBLE LOSSES, RESULTING FROM (A) YOUR ACCESS TO OR USE OF OR INABILITY TO ACCESS OR USE THE SITE; (B) ANY CONDUCT OR CONTENT OF ANY THIRD PARTY ON THE SITE, INCLUDING WITHOUT LIMITATION, ANY DEFAMATORY, OFFENSIVE OR ILLEGAL CONDUCT OF OTHER USERS OR THIRD PARTIES; OR (C) UNAUTHORIZED ACCESS, USE OR ALTERATION OF YOUR TRANSMISSIONS OR CONTENT. IN NO EVENT SHALL TRUTH INITIATIVE'S AGGREGATE LIABILITY FOR ALL CLAIMS RELATING TO THE SITE EXCEED ONE HUNDRED U.S. DOLLARS (U.S. \$100.00).

#### **Arbitration**

For any dispute you have with Truth Initiative regarding the Site shall be resolved by arbitration in accordance with the Commercial Arbitration Rules of the American Arbitration Association and judgment upon the arbitrator's award may be entered in any court having jurisdiction. The prevailing party in any such arbitration shall be entitled to recover reasonable attorney's fees from the other party. However, nothing shall prevent either you or Truth Initiative from seeking injunctive or other equitable relief from the courts for matters related to data security, intellectual property or unauthorized access to the Site. ANY AND ALL CLAIMS MUST BE BROUGHT IN THE PARTIES' INDIVIDUAL CAPACITY, AND NOT AS A PLAINTIFF OR CLASS MEMBER IN ANY PURPORTED CLASS OR REPRESENTATIVE PROCEEDING, AND, UNLESS BOTH PARTIES AGREE OTHERWISE, THE ARBITRATOR MAY NOT CONSOLIDATE MORE THAN ONE PERSON'S CLAIMS. YOU AGREE THAT, BY ENTERING INTO THESE TERMS, YOU AND TRUTH INITIATIVE ARE EACH WAIVING THE RIGHT TO A TRIAL BY JURY OR TO PARTICIPATE IN A CLASS ACTION.

### Governing Law and Jurisdiction

The Site is controlled and operated from the United States. These Terms shall be governed by the laws of the District of Columbia, without respect to its conflict of laws principles. You agree to submit to the personal jurisdiction of a local court located in the District of Columbia or the United States District Court for the District of Columbia, for any actions not subject to the arbitration provisions set forth above.

## **Indemnification and Hold Harmless**

You will indemnify and hold harmless Truth Initiative and its officers, directors, employees, and agents from any and all claims arising out of or related to (1) your Content and/or (2) your use of, or your inability to use, this Application or the information contained therein.

#### No Waiver

Truth Initiative's failure to assert any right or provision under these Terms shall not constitute a waiver of such right or provision.

# **Contacting Us**

If you have any questions about this Privacy Policy, Terms of Service or anything relating to the website, please contact us.